CLINICAL TRIAL: NCT01619553
Title: Identification of Genetic Variants That Contribute to Keloid Formation in Families and Isolated Cases.
Brief Title: Genetic Analysis of Keloids
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Ernst Reichenberger, Associate Professor, UConn Health
Other Study IDs: UCHC03-007
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Keloid
Keywords: keloid; fibrosis; wound healing; scar
MeSH Terms: conditions — Keloid; Fibrosis; Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, scar tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- affected: individuals with keloids
- unaffected: unrelated unaffected controls or unaffected family members

SUMMARY:
Keloids have a strong genetic component. The goal of this study is to identify genes and regulatory elements on chromosomes that are the cause for keloids or contribute to keloid scarring.

DETAILED DESCRIPTION:
Keloids are scars that keep growing beyond the border of the original wound. They typically persist for several years, expand for an extensive period of time and are sometimes called benign tumors. Keloids often have a lumpy surface and are often tender, itchy or inflamed around the growing border.

Keloids in most keloid patients do not run in the family. In the inheritable form of keloids it is possible that there is one major gene mutation that puts family members at risk for developing keloids. There may be other variations in the DNA (DNA makes up the chromosomes) that determine whether keloids become large and aggressive or stay small and without many symptoms.

For this study we will:

* Send out study participation kits and consent by phone
* Collect a saliva sample from eligible individuals
* Obtain information regarding the keloids
* Document keloids with photos
* If keloid patients undergo keloid surgery we ask to obtain some scar tissue that would otherwise be discarded
* Isolate DNA from the saliva sample
* Perform genetic analyses of the DNA with the most up-to-date methods available to identify genetic variations
* Study in the laboratory why the genetic variations cause keloids

ELIGIBILITY:
Inclusion Criteria:

* keloids;
* unaffected individuals only if part of a participating keloid family

Exclusion Criteria:

* no keloids;
* unaffected individuals only as part of a participating keloid family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with diagnosed keloids.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2009-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic elements | at time of identification
  The goal is to identify relevant genes or genetic elements that cause the disease or contribute to the disease progression and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Reichenberger, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center (UCHC), Farmington, Connecticut, United States

REFERENCES:
- [Background] Marneros AG, Norris JE, Watanabe S, Reichenberger E, Olsen BR. Genome scans provide evidence for keloid susceptibility loci on chromosomes 2q23 and 7p11. J Invest Dermatol. 2004 May;122(5):1126-32. doi: 10.1111/j.0022-202X.2004.22327.x. PMID 15140214
- [Background] Marneros AG, Norris JE, Olsen BR, Reichenberger E. Clinical genetics of familial keloids. Arch Dermatol. 2001 Nov;137(11):1429-34. doi: 10.1001/archderm.137.11.1429. PMID 11708945
- [Background] Santos-Cortez RLP, Hu Y, Sun F, Benahmed-Miniuk F, Tao J, Kanaujiya JK, Ademola S, Fadiora S, Odesina V, Nickerson DA, Bamshad MJ, Olaitan PB, Oluwatosin OM, Leal SM, Reichenberger EJ. Identification of ASAH1 as a susceptibility gene for familial keloids. Eur J Hum Genet. 2017 Oct;25(10):1155-1161. doi: 10.1038/ejhg.2017.121. Epub 2017 Jul 26. PMID 28905881
- See also: Reichenberger lab research information — https://health.uconn.edu/reichenberger-lab/